CLINICAL TRIAL: NCT02618382
Title: A Study on the Safety of Tranexamic Acid for the Chronic Subdural Hematoma Population
Acronym: TXA in CSDH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Collaborators: Barrow Neurological Foundation (Other)
Responsible Party: Principal Investigator, Lisa Arnold, Research manager, St. Joseph's Hospital and Medical Center, Phoenix
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHX15BN048
Record Dates: First submitted 2015-11-23; First posted 2015-12-01 (Estimated); Results first posted 2021-11-09 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Subdural Hematoma
MeSH Terms: conditions — Hematoma, Subdural | interventions — Tranexamic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All subjects (Experimental): Patients will undergo standard treatment of their chronic subdural hematoma with the addition of preoperative and postoperative oral tranexamic acid treatment. Patients will receive a dose of 1300mg orally three to four hours prior to surgery. They will then take 1300mg orally three times daily for three days or until discharge, whichever occurs first.
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid — 1300mg tranexamic acid by mouth once before surgery and then three times a day for up to three days or until they are discharged from the hospital, whichever comes first
  Other Names: Lysteda; Cyklokapron

SUMMARY:
This is a single center single arm study of 50 patients to 1) determine the safety of tranexamic acid in the chronic subdural hematoma population following surgical drainage of chronic subdural hematomas and 2) determine if the use of oral tranexamic acid reduces the rate of ipsilateral recurrence following drainage of chronic subdural hematomas. This will be compared to historical controls. This study intends to be a prerequisite to a large nationally funded randomized control trial.

DETAILED DESCRIPTION:
Chronic subdural hematomas are a common problem faced by neurosurgery with an annual incidence of 13.5/100,00 persons per year and up to 58/100,000 in the over 65 years old population. Their treatment is often complicated by recurrence with rates reported as high as 33%. Currently there is no good strategy to help avoid this problem, which adds significantly to patient morbidity. The pathogenesis of this problem is believed to be related to the propensity of the associated neo-membranes to bleed. It has been shown with labeled red blood cells that bleeding continues to occur into the hematoma cavity. It has also been shown that there are high levels of tissue plasminogen activator in the outer membrane of chronic subdural hematomas. It has been found that ratio of tissue plasminogen activator to plasminogen activator inhibitor contributed to the pathogenesis. It has also been shown that chronic subdural hematomas have high levels of fibrin degradation products which in addition to marking the breakdown of fibrin are themselves antihemostatic by enhancing tissue plasminogen activator activity, having an antithrombin affect and inhibiting platelet aggregation and fibrin polymerization. Essentially, a scenario of ongoing hemorrhage and repeated clot formation and hyperfibrinolysis leads to the expansion and recurrence of chronic subdural hematomas.

Given the importance of plasmin and hyperfibrinolysis in the pathophysiology of chronic subdural hematomas, interrupting its action and the vicious cycle it propagates seems an ideal therapeutic target. Tranexamic acid is a synthetic lysine amino acid derivative. It binds to the fibrin binding sites on plasmin or plasminogen and prevents its interaction and degradation of fibrin. This effect on the neo-membranes of chronic subdural hematomas should prevent rebleeding and the reaccumulation of the subdural hematoma.

Tranexamic acid has been shown to be safe and effective in reducing blood loss and transfusions in a number of types of surgery, reduced mortality and need for urgent surgery in patients with GI bleeding, and reduced bleeding associated with menorrhagia and pregnancy. Adverse effects are generally mild. Thought there is a theoretical increased risk of thromboembolic complications, multiple randomized controlled trials have not shown an increased risk. Furthermore, in a study of over 3000 gynecologic patients using tranexamic acid, there were no thromboembolic complications. This is likely because tranexamic acid has been shown to not have an effect on plasminogen in the vein wall.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing intervention for chronic subdural hematoma (cSDH) including drainage
* cSDH will be defined as hematoma on CT imaging that is predominantly iso- to hypodense to brain
* 18-85 years of age

Exclusion Criteria:

* cSDH not requiring surgical drainage
* patients undergoing bedside twist drill craniostomy
* medically unstable for surgery
* patients requiring long-term anticoagulation (unable to stay off for less than 30 days)
* patients not expected to survive to the completion of followup
* patients comatose prior to the initiation of treatment
* history of thromboembolic problem including stroke, myocardial infarction, deep vein thrombosis and/or pulmonary embolism
* pregnant
* minor
* allergy/sensitivity to tranexamic acid
* irreversible coagulopathy
* known clotting disorder
* bilateral hematomas with both requiring drainage
* incarcerated
* any patient not judged suitable for the study by the investigators
* women who are taking combination hormonal contraception

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2018-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew S Little, MD, Principal Investigator — Barrow Brain and Spine, Phoenix, AZ
Locations (1):
- Barrow Brain and Spine, Phoenix, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from a single major neurological center from Nov 2015 to Aug 2017. Patients between the ages 18 and 85 undergoing operative treatment with postop drainage of chronic SDH were evaluated for inclusion. Participants received a single dose of tranexamic acid 1300 mg preop and then 3 times daily for 3 days postop or until dc
Period: Overall Study
Arm/Group | All Subjects
Started | 32 (Enrolled and consented for study treatment)
Completed | 29 (Completed Study treatment)
Not Completed | 3
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Subjects
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 17
Age, Continuous [Mean (Full Range); unit: years] | 66 [40 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 21
  More than one race | 06
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Medication Related (Thromboembolic) Complications
Description: occurrence of stroke, myocardial infarction, deep vein thrombosis, and/or pulmonary embolism within 30 days
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | All Subjects
Number analyzed (Participants) | 32
Participants | 0

2. Secondary Outcome: Hematoma Thickness on CT Scan
Description: Hematoma width (measured in cm) on post operative CT scans compared to baseline (preoperative). Preoperative axial non-contrast CT images were reviewed by a study investigator for maximal hematoma thickness, the presence of septations, and midline shift. Septations were determined to be present if there were thin, hyperdense, dividing membranes within the limits of the subdural collection. Postoperative axial non-contrast CT was planned within 24 hours post surgery and on postoperative days 3 and 30 (which could be scheduled within 7 days of the 30-day mark) to determine maximal hematoma thickness and midline shift using the preoperative methodology.
Time Frame: postoperative days 1, 3, and 30+/-7 days
Population: 1 participant did not receive 3-day post-operative follow-up CT because they were discharged home prior to day 3.
  8 participants did not receive 30-day postoperative follow-up CT: in 5 of these patients, postoperative imaging was deemed unnecessary by the treating provider because of the patients' clinical progress. In the other 3 patients, follow-up imaging was obtained with magnetic resonance imaging rather than CT, as dictated by the treating surgeon
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | All Subjects
Number analyzed (Participants) | 32
centimeters
  Preop (Baseline) hematoma thickness | 2.24 (0.65)
  Postop day 1 - hematoma thickness | 1.17 (0.53)
  Postop day 3 - hematoma thickness: number analyzed (Participants) | 31
  Postop day 3 - hematoma thickness | 1.28 (0.55)
  Postop day 30 - hematoma hematoma thickness: number analyzed (Participants) | 24
  Postop day 30 - hematoma hematoma thickness | 0.73 (0.73)
Statistical Analysis 1: Comparison: All Subjects; Nonparametric tests were used for statistical comparison, including the Kruskal-Wallis rank-sum test for multiple groups and the Mann-Whitney U test for 2 groups. P values <0.05 were considered statistically significant. Data tabulation and analysis were performed using R statistical software version 3.4.2 (R Foundation for Statistical Computing, Vienna, Austria); Test type: Superiority; p < 0.05, ANOVA — The P values for differences among time point means were determined by ANOVA for continuous variables

3. Secondary Outcome: Functional Status Determined by Modified Rankin Score (mRS) From Baseline to 30 Days Postop
Description: The Modified Rankin Score (mRS) is a 6 point disability scale with scores ranging from 0 to 5. A separate category of 6 is usually added for patients who expire.
  Lower score of 0, 1,2 are the best outcome up to 5 with worst outcome. 0 The patient has no residual symptoms.
  1. The patient has no significant disability; able to resume all pre-stroke activities.
  2. The patient has slight disability; unable to resume all pre-stroke activities but able to look after self without daily help.
  3. The patient has moderate disability; requiring some external help but able to walk without the assistance of another individual.
  4. The patient has moderately severe disability; unable to walk or attend to bodily functions without assistance.
  5. The patient has severe disability; bedridden, incontinent, requires continuous care.
  6. The patient has expired (during the hospital stay or after discharge from the hospital).
  A chi -squared test was used for categorical value
Time Frame: Measured between 2 timepoints: Baseline(Day 0) and postoperative (day 30)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Subjects
Number analyzed (Participants) | 32
score on a scale
  Baseline mRS Score | 2.3 (1.3)
  Postop Day 30 mRS score | 0.9 (1.1)
Statistical Analysis 1: Comparison: All Subjects; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.05, ANOVA — Paired comparison of hematoma thickness at defined time point means determined by ANOVA for continuous variables

4. Secondary Outcome: Change in National Institute of Health Stroke Scale (NIHSS)
Description: National Institute of Health Stroke Scale (NIHSS) (0-42); 0 is better, 42 is worse.
  The NIHSS measures several aspects of brain function, including consciousness, vision, sensation, movement, speech, and language. A certain number of points are given for each of these physical and cognitive functions during a focused neurological examination. A maximum score of 42 represents the most severe and devastating stroke.
  The levels of stroke severity as measured by the NIHSS scoring system are:
  0 = no stroke 1-4 = minor stroke 5-15 = moderate stroke 15-20 = moderate/severe stroke 21-42 = severe stroke
Time Frame: Immediately preoperative (Day 0) and discharge (up to 30 days postoperative)
Population: NIHSS Assessment was not done at postoperative day 30 secondary to non in person visit. Other assessments for these 4 participants were done via telephone.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Subjects
Number analyzed (Participants) | 32
score on a scale
  Preop (baseline) NIHSS Score | 1.7 (1.5)
  Postop day 30 NIHSS Score: number analyzed (Participants) | 28
  Postop day 30 NIHSS Score | 0.2 (0.4)
Statistical Analysis 1: Comparison: All Subjects; [analysis description as in outcome 2, analysis 1]; Test type: Other; p < 0.05, ANOVA — The P values for differences among time point means were determined by ANOVA for continuous variables and by chi-squared test for categorical values in grouped mRS scores

ADVERSE EVENTS:
Time Frame: at 30 days
Arm/Group | All Subjects
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 7/32
Other Adverse Events (participants affected / at risk) | 7/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=32)
Wound infection (Infections and infestations) | 3 (3) — infection at site of surgical wound
Alcohol withdrawal syndrome (Psychiatric disorders) | 2 (2) — Delirium tremors from alcohol withdrawal
Epidural hemorrhage (Vascular disorders) | 1 (1) — spontaneous epidural hemorrhage
seizure (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=32)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1) — Disturbances in consciousness, NEC
hyponatremia (Metabolism and nutrition disorders) | 5 (5) — sodium less < 135 mmol/L

LIMITATIONS AND CAVEATS:
This study limitations include its small size, lack of a control group, and deviations in study protocol with regard to postoperative imaging. Given that the study was not designed to determine the relative effectiveness of TXA in preventing recurrence, factors that may have influenced the recurrence rate, such as hematoma size, hematoma characteristics, and surgical technique, were unable to be controlled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-09): https://cdn.clinicaltrials.gov/large-docs/82/NCT02618382/Prot_SAP_000.pdf